CLINICAL TRIAL: NCT01113411
Title: Effectiveness of Intensive Rehabilitation on Shoulder Function After a Fracture of the Proximal Humerus Treated by Locked Plate. A Prospective Randomized Study
Brief Title: Effectiveness of Intensive Rehabilitation on Shoulder Function After Proximal Humerus Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hopital de l'Enfant-Jesus (Other)
Responsible Party: Principal Investigator, Pelet Stephane, Dr Stephane Pelet MD, PhD Orthopedic surgeon, Hopital de l'Enfant-Jesus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEJ-525
Record Dates: First submitted 2010-04-28; First posted 2010-04-29 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Fracture of Proximal Humerus
Keywords: humerus fracture; locked plate
MeSH Terms: conditions — Humeral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive Rehabilitation (Active Comparator)
  Interventions: Device: PHILOS™ locked plate system by Synthes Canada©; Other: Early and intensive exercise program
- Standard Rehabilitation (Active Comparator)
  Interventions: Device: PHILOS™ locked plate system by Synthes Canada©; Other: Standard rehabilitation program

INTERVENTIONS:
Device: PHILOS™ locked plate system by Synthes Canada© — The surgery will be performed under standardized general anesthetic with a prophylactic antibiotic. The deltopectoral approach is used in all cases. The fracture will be fixed using the PHILOS locked plate system by Synthes Canada ©. Some additional osteosutures may be used. The wound is irrigated and then closed in two layers at the end of intervention. A splint thoracic brace will be installed in all patients before the end of anesthesia.
Other: Early and intensive exercise program — A thoraco brachial brace will be worn for 48 hours following the surgery and then removed for the remainder of treatment. Patients will then start the intensive rehabilitation program without physical therapy. The exercise program will be provided to the patient.
  The exercises consist of active and active assisted movements of the shoulder for a period of six weeks, limiting external rotation to 0 °. Patients are encouraged to use their affected limb for daily activities. Strengthening exercises are started the 6th week following surgery and the full program will be completed three months after surgery. Patients who wish can then continue their rehabilitation with a physiotherapist.
  The patient will complete a daily diary to validate the frequency and intensity of the exercises.
  Arms: Intensive Rehabilitation
Other: Standard rehabilitation program — The patient will wear the thoraco brachial brace for a period of four weeks following the surgery. It may be taken off for hygiene purposes and dressing up. After the four weeks, the patient will take the brace off permanently and begins an exercise program, writing down the frequency and intensity of the exercises. Physiotherapy is allowed for the remaining part of the three months rehabilitation program.
  Arms: Standard Rehabilitation

SUMMARY:
The fracture of the proximal humerus represents 4% of the fractures encountered in clinics and it must be treated surgically. Thus, the aim of the surgical treatment is to maintain bone alignment, articular congruity, vascularization of the humeral head and provide a painless shoulder with satisfactory function.

The objective of this study is to demonstrate the potential benefits of an early rehabilitation program on shoulder function.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years
* Unstable fracture of the proximal humerus
* Two-part and three-part fractures according to the Neer classification
* Closed fracture
* Time between trauma and surgery less than or equal to 7 days
* Signing of consent form

Exclusion Criteria:

* Stable fracture of the proximal humerus (not requiring surgery)
* Four-part fracture on the Neer classification
* Fracture-dislocation or fracture involving the articular surface
* Isolated fracture of the large or small tuberosity
* Pathological fracture
* Fracture associated with neuro-vascular lesions
* Bilateral fractures
* Fracture associated with long bones fracture
* Polytrauma
* Previous history of fracture or surgery to the ipsilateral proximal humerus
* Severe COPD
* Severe neuromuscular disorders (Parkinson, hemiparesis, myasthenia gravis, muscular dystrophy, etc. ...)
* Remote location of patient's home which makes it difficult to come to facility for follow-up visits
* Any medical condition making it impossible for the patient to perform the exercise program (Alzheimer, dementia, etc. ...)
* Man or woman incapacitated sign consent form
* Any other condition which prevents the assessor from fully monitoring the patient during study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Functional outcome on Constant score | 6 months after surgery
  The investigators will validate that early and intensive rehabilitation gives a better functional outcome at 6 months using the Constant score adjusted for age. A difference of 10 points is considered significant (standard deviation of 15 points).

SECONDARY OUTCOMES:
Proportion of reoperation | within the first year following surgery
  The rate of complications such as infection, implant removal, implant failure and necrosis which necessitate additional surgery.
Loss of radiological reduction | 1 or 2 days after surgery
  The main displacements occur in varus and it will be measured on a radiography on an AP view of Neer. The neck-shaft angle will be measured and a difference of 10 degrees will be considered significant to account for the lack of standardization of the radiological technique.
Loss of radiological reduction | 10-14 days after surgery
  The main displacements occur in varus and it will be measured on a radiography on an AP view of Neer. The neck-shaft angle will be measured and a difference of 10 degrees will be considered significant to account for the lack of standardization of the radiological technique
Loss of radiological reduction | 3 or 4 months after surgery
  The main displacements occur in varus and it will be measured on a radiography on an AP view of Neer. The neck-shaft angle will be measured and a difference of 10 degrees will be considered significant to account for the lack of standardization of the radiological technique
Loss of radiological reduction | 6 months after surgery
  The main displacements occur in varus and it will be measured on a radiography on an AP view of Neer. The neck-shaft angle will be measured and a difference of 10 degrees will be considered significant to account for the lack of standardization of the radiological technique
Loss of radiological reduction | 12 months after surgery
  The main displacements occur in varus and it will be measured on a radiography on an AP view of Neer. The neck-shaft angle will be measured and a difference of 10 degrees will be considered significant to account for the lack of standardization of the radiological technique
Sustainability of the efficacy on Constant score | 12 months after surgery
  Constant score will be measured one year after surgery to demonstrate the sustainability of the efficacy of intensive rehabilitation.
Quality of life on DASH scale | 3 months after surgery
  The quality of life is measured using the DASH scale 3 months after surgery.
Quality of life on DASH scale | 6 months after surgery
  Quality of life is measured using the DASH scale 6 months after surgery.
Quality of life on DASH scale | 12 months after surgery
  Quality of life is measured using the DASH scale 12 months after surgery.
Return to professional activities | 3 or 4 months after surgery
  This will be determined in days after surgery, to rates of 50% and 100% of the usual workload.
Pain on visual analog scale (VAS) | 10-14 days after surgery
  The measure will be carried out using a suitable rule designed for this type of measurement, counting only full numbers from 1 to 10 on VAS.
Pain on VAS | 3 or 4 months after surgery
  The measure will be carried out using a suitable rule designed for this type of measurement, counting only full numbers from 1 to 10 on VAS.
Pain on VAS | 6 months after surgery
  The measure will be carried out using a suitable rule designed for this type of measurement, counting only full numbers from 1 to 10 on VAS.
Pain on VAS | 12 months after surgery
  The measure will be carried out using a suitable rule designed for this type of measurement, counting only full numbers from 1 to 10 on VAS.
Measurement of range of motion of shoulder | 3 months after surgery
  Using a goniometer, we will measure the bending (normal value 180 °), abduction (180 °), external rotation in the scapular plane (90 °) and internal rotation in the plane scapula (60 °).
Measurement of range of motion of shoulder | 6 months after surgery
  Using a goniometer, we will measure the bending (normal value 180 °), abduction (180 °), external rotation in the scapular plane (90 °) and internal rotation in the plane scapula (60 °).
Measurement of range of motion of shoulder | 12 months after surgery
  Using a goniometer, we will measure the bending (normal value 180 °), abduction (180 °), external rotation in the scapular plane (90 °) and internal rotation in the plane scapula (60 °).

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Pelet, MD, PhD, Principal Investigator — Hôpital Enfant-Jésus; Annie Arteau, MD, Principal Investigator — Hôpital Enfant-Jésus
Locations (1):
- CHA-Pavillon Enfant-Jésus, Québec, Quebec, Canada

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196